CLINICAL TRIAL: NCT06532981
Title: The Effect of the Ankle-foot Orthosis on Muscle Activity in the Lower Limbs in Children With Cerebral Palsy
Brief Title: The Effect of AFOs on the EMG of Children With CP
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s65337_s66532_EMG
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral Palsy; Rehabilitation; Gait analysis; Variability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory children with spastic CP: Ambulant children with cerebral palsy between 6 and 17 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.

SUMMARY:
Children with cerebral palsy (CP) have altered gait patterns as a result of primary and secondary symptoms. Ankle-foot orthoses (AFOs) are frequently used to improve their gait. Despite evidence of AFO-effects on gait kinetics and -kinematics, the effects on muscle activity remain unclear.

This study will investigate the effect of AFOs on the amplitude and timing, as well as the co-activation of lower limb muscle activity in children with spastic CP.

DETAILED DESCRIPTION:
With a prevalence of two to three per 1000 live births, Cerebral Palsy (CP) is the most common motor disability of childhood. Improving disturbed gait in ambulatory children with CP is an important treatment goal because it is associated with functional independence and participation of children in the society. It is a common practice to prescribe ankle-foot orthoses (AFO) for ambulatory children to improve their gait, prevent secondary deformities, provide an improved base of support, and compensate for muscle weakness.

Previous research highlighted that there is a direct effect on the muscle activity of the distal muscles and an indirect effect on the proximal muscles. However, the impact of the AFO on the muscle activity of the plantar and dorsiflexors is clinically relevant since reduced muscle activity may lead to muscle atrophy and altered motor control. Therefore, more research is needed on the effect of AFOs on the medial gastrocnemius and the tibialis anterior, in both unilaterally and bilaterally involved children. Moreover, the impact of the AFO on the muscle activity of the quadriceps, apart from the hamstrings, needs to be further explored as well.

The purpose of the current study is to investigate the effect of the AFO on muscle activity in the distal and proximal leg muscles of children with CP while walking.

On the measurement day, subjects will first receive a standard clinical examination preceding the clinical overground three-dimensional gait analysis (3DGA) that is planned as a routine clinical follow-up at the CMAL (clinical motion analysis laboratory), extended with an additional 3DGA on the treadmill. The treadmill gait laboratory and overground gait laboratory are across the hall from each other, which makes it possible for the subject to walk from one to the other gait laboratory in just a minute. During the 3DGA, kinematic, kinetic and EMG-data will be collected.

ELIGIBILITY:
Inclusion criteria:

* Gross Motor Function Classification System (GMFCS) level I - III
* CP (bilateral & unilateral)
* Age: 6 - 17 years
* Prescribed AFO by the medical team (as part of the standard care)

Exclusion criteria:

* Severe contractures or spasticity, which makes it impossible to wear a conventional AFO
* Cognitive or visual impairment that hinder them to understand instructions
* Previous surgery on bones and/or muscles of the legs in the last 12 months prior to assessment
* Presence of ataxia or dystonia

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ambulant children with cerebral palsy between 6 and 17 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EMG-waveform amplitude & timing | One measurement of 150 minutes
  The averaged time-normalized continuous EMG-waveforms for each walking condition (i.e., barefoot, AFO, overground and on the treadmill) the following muscles: the quadriceps (m. rectus femoris, m. vastus lateralis), the hamstrings (m. semitendinosus, m. biceps femoris) and the shank (m. gastrocnemius medialis, m. tibialis anterior).
EMG co-activation | One measurement of 150 minutes
  The co-activation was calculated by defining the synchronised activations of the agonist and antagonist muscles. To quantify the co-activation, the on- and off-timing of the muscle activity needed to be defined for the rectus femoris, the medial hamstrings, the gastrocnemius and the tibialis anterior.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium